CLINICAL TRIAL: NCT01391585
Title: Expanding Comparative Effectiveness Research (CER) Capability Through Complex Patient Relationship Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Henry Fischer, MD, Denver Health and Hospital Authority
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R24HS019453-01PRM; R24HS019453-01 (NIH)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes; Hyperlipidemia
Keywords: Text; SMS; diabetes; self-monitoring; self-management; adherence
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- text message recipients (Experimental): Patients will be recruited to receive text messages
  Interventions: Other: Text Message prompts

INTERVENTIONS:
Other: Text Message prompts — In this single armed intervention, patients will receive text message prompts

SUMMARY:
The investigators are testing whether patients with diabetes can communicate with our health care system through text messaging. The investigators will look at how often they respond to prompts for blood pressures, blood sugars, and step counts. The investigators will also see if they come in for lab tests when prompted by text message. Also, for patients overdue for medication refills, the investigators will ask them why they have not yet called for the refill.

DETAILED DESCRIPTION:
Patients will be sent text messages through a software interface, the Patient Relationship Manager (PRM). A registered nurse will also use PRM to receive incoming responses. Tasks will be created for her to outreach to patients who have out of range text responses or poor response rates. This intervention if a feasibility study to see if patients can communicate with the investigator's health care system and potentially utilize PRM to better manage their diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* diabetes
* own a cell phone
* 2 primary care visits in last year
* English or Spanish speaking

Exclusion Criteria:

* End-stage disease with estimate of less than 6 months to live

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
response rate to home monitoring prompts | 4 months
  resonse rate to blood pressure, blood sugar, and step count prompts

SECONDARY OUTCOMES:
response rate to prompt for lab text by text message | 4 months
  response rate to prompt for lab text by text message
response to barrier questions for non-adherence | 4 months
  We will analyze the responses to text message prompts in patients late for picking up medications.

CONTACTS AND LOCATIONS:
Overall Officials: henry h fischer, MD, Principal Investigator — Denver Health
Locations (1):
- Denver Health, Denver, Colorado, United States